CLINICAL TRIAL: NCT03404960
Title: PARPVAX: Parpvax: A Phase 1b/2, Open Label Study of Niraparib Plus Either Ipilimumab or Nivolumab in Patients With Advanced Pancreatic Cancer Whose Disease Has Not Progressed on Platinum-based Therapy
Brief Title: Niraparib + Ipilimumab or Nivolumab in Progression Free Pancreatic Adenocarcinoma After Platinum-Based Chemotherapy
Acronym: Parpvax
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Bristol-Myers Squibb (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 828516
Record Dates: First submitted 2017-12-19; First posted 2018-01-19 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Platinum; chemotherapy; Niraparib; Ipilimumab; Nivolumab; Pancreatic adenocarcinoma; PARP inhibitor; Pancreatic ductal adenocarcinoma; DDR; PDAC
MeSH Terms: interventions — niraparib; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Niraparib + Nivolumab
  Interventions: Drug: Niraparib + Nivolumab
- Arm B (Experimental): Niraparib + Ipilimumab
  Interventions: Drug: Niraparib + Ipilimumab

INTERVENTIONS:
Drug: Niraparib + Nivolumab — Niraparib 200mg PO daily on days 1-28 of each 28-day cycle. Nivolumab 480mg IV day 1 of each cycle.
  Other Names: Arm A
  Arms: Arm A
Drug: Niraparib + Ipilimumab — Niraparib 200mg PO daily on days 1-21 of each 21-day cycle. Ipilimumab 3mg/kg IV day 1 of each cycle, for the first 4 cycles only.
  Other Names: Arm B
  Arms: Arm B

SUMMARY:
The main purpose of this study is to look at the effectiveness, safety, and anti-tumor activity (preventing growth of the tumor) of the drugs Niraparib with either Ipilimumab or Nivolumab on patients and their pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma with locally advanced or metastatic disease
2. ≥18 years of age
3. Patients must be able to understand the study procedures and agree to participate in the study by providing written informed consent
4. Patients must have received treatment with platinum-based (cisplatin, oxaliplatin or carboplatin) treatment for locally advanced or metastatic pancreatic cancer and have received a minimum of 16 weeks of therapy without evidence of disease progression based on the investigator's opinion. This does not have to be the patient's current treatment.

   * This requires at least stable imaging and a stable or decreasing tumor marker as applicable and as determined by the investigator.
   * If a patient has demonstrated a biochemical and imaging response to platinum therapy and has not progressed within 16 weeks of starting this therapy but had to discontinue platinum prior to 16 weeks for a legitimate medical reason (as determined by the investigator), the patient may still be considered for the trial
5. Patients may have previously failed non-platinum containing therapy or may never have previously progressed on treatment

   * Discontinuation of the platinum component of the regimen for chemotherapy-related toxicity is permissible provided the patient has previously received at least 16 weeks of platinum-based therapy without evidence of disease progression ≤8 weeks after treatment with the platinum agent
6. Measurable disease is not a requirement for study entry
7. Female participant has a negative serum pregnancy test within 24 hours prior to taking study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 6 months after the last dose of study treatment, or is of nonchildbearing potential
8. Male patient agrees to use an adequate method of contraception starting with the first dose through 90 days after the last dose of study treatment
9. Adequate organ function confirmed by the following laboratory values obtained ≤7 days prior to the first day of study therapy:

   * Absolute neutrophil count (ANC) ≥1.5 x 109/L
   * Platelets>100 x 109/L
   * Hemoglobin ≥9g/dL
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 x upper limit of normal (ULN); if liver metastases, then ≤5 x ULN
   * Total bilirubin ≤1.5 x ULN; if liver metastases or metabolic disorder such as Gilbert's syndrome, then ≤2.5 x ULN.
   * Serum creatinine ≤1.5 x ULN or estimated glomerular filtration rate (GFR) ≥45 mL/min using Cockcroft Gault formula.
10. Eastern Cooperative Oncology (ECOG) performance status of 0 to 1.

Exclusion Criteria:

1. Prior treatment with a PARP inhibitor, ipilimumab, nivolumab or other cytotoxic T-lymphocyte-associated protein (CTLA-4), PD-1 or PD-L1 inhibitor.
2. Patients who have demonstrated resistance to platinum agents (e.g. oxaliplatin, cisplatin) are not eligible to participate in this study
3. Clinical evidence of uncontrolled malabsorption and/or any other gastrointestinal disorder or defect that would, in the opinion of the investigator, interfere with the absorption of niraparib
4. Acute infection requiring intravenous antibiotics, antiviral or antifungal agents during the 14 days prior to first dose of study therapy
5. Patients will be excluded if they have an active, known or suspected autoimmune disease, defined as: patients with a history of inflammatory bowel disease are excluded from this study, as are patients with a history of symptomatic autoimmune disease (e.g. rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus, autoimmune vasculitis e.g. Wegener's Granulomatosis); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome).

   NOTE: Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
6. Has a history of interstitial lung disease or active, non-infectious pneumonitis
7. Has received a live vaccine within 4 weeks prior to the first dose of trial therapy (Note: seasonal influenza vaccines for injection are generally inactivated and are allowed; however intranasal influenza vaccines (e.g. Flu-Mist) are live attenuated vaccines and are not allowed
8. For fertile patient (female able to become pregnant or male able to father a child), refusal to use effective contraception during the period of the trial and:

   * Female patients refusing to use effective contraception for 6 months after the last dose of study drug.
   * Male patients refusing to use effective contraception for 90 days after the last dose of study drug.
9. Received any systemic treatment for pancreatic cancer ≤14 days prior to first dose of therapy. Patients must not have had investigational therapy administered ≤4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is longer, prior to the first scheduled day of dosing in this study
10. Patients will be excluded if they have a condition requiring systemic treatment with either corticosteroids (>10mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses >10mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
11. Patient has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
12. Non-study related minor surgical procedure ≤5 days, or major surgical procedure ≤21 days, prior to the first dose of therapy; in all cases, patients must be sufficiently recovered and stable before treatment administration.
13. Active drug or alcohol use or dependence that would interfere with study compliance.
14. Presence of any other condition that may increase the risk associated with study participation or may interfere with the interpretation of study results, and, in the opinion of the investigator, would make the patient inappropriate for entry into the study.
15. Patient must not have any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
16. Patients must not be simultaneously enrolled in any therapeutic clinical trial
17. Patients must not have had radiotherapy within 4 weeks of the first dose of study treatment
18. Patients must not have a known hypersensitivity to the components of niraparib or the excipients
19. Patients must not have received a transfusion (platelets or red blood cells) ≤ 4 weeks of the first dose of study treatment
20. Patients must not be undergoing treatment for an active cancer at the time of randomization. Exceptions include: local therapies for skin cancers and hormonal therapies for breast or prostate cancer.
21. Patients must not have a history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS), and must not test positive for HIV during study screening.
22. Patients must not have known, symptomatic brain or leptomeningeal metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2024-10-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Reiss KA, Mick R, Teitelbaum U, O'Hara M, Schneider C, Massa R, Karasic T, Tondon R, Onyiah C, Gosselin MK, Donze A, Domchek SM, Vonderheide RH. Niraparib plus nivolumab or niraparib plus ipilimumab in patients with platinum-sensitive advanced pancreatic cancer: a randomised, phase 1b/2 trial. Lancet Oncol. 2022 Aug;23(8):1009-1020. doi: 10.1016/S1470-2045(22)00369-2. Epub 2022 Jul 7. PMID 35810751

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 104 subjects enrolled. 11 failed eligibility criteria. 2 withdrew consent. 91 randomly assigned and included in the safety analysis.
Groups:
- Niraparib + Nivolumab (Arm A): Niraparib + Nivolumab: Niraparib 200mg PO daily on days 1-28 of each 28-day cycle.
  Nivolumab 480mg IV day 1 of each cycle.
- Niraparib + Ipilimumab (Arm B): Niraparib + Ipilimumab: Niraparib 200mg PO daily on days 1-21 of each 21-day cycle.
  Ipilimumab 3mg/kg IV day 1 of each cycle, for the first 4 cycles only.
Period: Overall Study
Arm/Group | Niraparib + Nivolumab (Arm A) | Niraparib + Ipilimumab (Arm B)
Started | 46 | 45
Completed | 44 | 40
Not Completed | 2 | 5
Not completed — Adverse Event | 0 | 2
Not completed — Rapidly declined before 1st follow-up scan | 0 | 2
Not completed — Bowel obstruction | 0 | 1
Not completed — Incorrect pathological diagnosis on internal review | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Niraparib + Nivolumab
  Niraparib + Nivolumab: Niraparib 200mg PO daily on days 1-28 of each 28-day cycle.
  Nivolumab 480mg IV day 1 of each cycle.
- Arm B: Niraparib + Ipilimumab
  Niraparib + Ipilimumab: Niraparib 200mg PO daily on days 1-21 of each 21-day cycle.
  Ipilimumab 3mg/kg IV day 1 of each cycle, for the first 4 cycles only.
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 44 | 40 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 23 | 41
  >=65 years | 26 | 17 | 43
Age, Continuous [Median (Full Range); unit: years] | 68 [46 to 84] | 64 [48 to 81] | 66 [46 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 20 | 35
  Male | 29 | 20 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 38 | 37 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 44 | 40 | 84

OUTCOME MEASURES:

1. Primary Outcome: Rate of Progression-free Survival at 6 Months (PFS6)
Description: The PFS6 rate will be estimated using the Kaplan-Meier method, and the 95% confidence interval will be estimated from the Kaplan-Meier curve. The null hypothesis is that the PFS6 rate in this population of subjects is 44%.
  Progressive disease is defined as at least a 20% increase in the sum of all the longest diameter (LD) of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. The appearance of one or more new lesions is also considered progression.
  Target lesions assessed according to RECIST v1.1.
Time Frame: 6 months after initiation of study therapy
Population: The efficacy population will consist of all patients who received at least one dose of study treatment and had a least one post-treatment assessment of response by RECIST v.1.1.
Measure: Number (95% Confidence Interval); unit: percentage of participants with PFS
Arm/Group | Niraparib + Nivolumab (Arm A) | Niraparib + Ipilimumab (Arm B)
Number analyzed (Participants) | 44 | 40
percentage of participants with PFS | 20.6 [8.3 to 32.9] | 59.6 [44.3 to 74.9]

2. Secondary Outcome: Objective Response Rate (ORR) Per RECIST v.1.1 as Assessed by Radiology Review
Description: The proportion of patients who achieve a complete or partial response, as determined by RECIST
Time Frame: From first restaging assessment through completion of study treatment (maximum 42 months)
Population: The efficacy population consisted of all patients who received at least one dose of study treatment and had at least one post-treatment assessment of response by RECIST.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Niraparib + Nivolumab (Arm A): Niraparib 200mg PO daily on days 1-28 of each 28-day cycle. Nivolumab 480mg IV day 1 of each cycle.
- Niraparib + Ipilimumab (Arm B): Niraparib 200mg PO daily on days 1-21 of each 21-day cycle. Ipilimumab 3mg/kg IV day 1 of each cycle, for the first 4 cycles only.
Arm/Group | Niraparib + Nivolumab (Arm A) | Niraparib + Ipilimumab (Arm B)
Number analyzed (Participants) | 44 | 40
Percentage of participants | 7.7 [1.5 to 19.5] | 15.4 [5.9 to 30.5]

3. Secondary Outcome: Overall Survival (OS)
Description: Start of treatment to death due to any cause or last patient contact alive.
Time Frame: Cycle 1 Day 1 until death, loss to follow-up, withdrawal of consent or until 5 years have passed, whichever occurs first
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Niraparib + Nivolumab (Arm A) | Niraparib + Ipilimumab (Arm B)
Number analyzed (Participants) | 44 | 40
Months | 13.2 [8.1 to 16.7] | 17.3 [12.8 to 21.9]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from 6 months after initiation of study therapy. All-Cause Mortality was from Cycle 1 Day 1 until death, loss to follow-up, withdrawal of consent or until 5 years have passed, whichever occurs first.
Description: The safety population consisted of all patients who received at least one dose of study treatment.
Arm/Group | Niraparib + Nivolumab (Arm A) | Niraparib + Ipilimumab (Arm B)
All-Cause Mortality (participants affected / at risk) | 7/46 | 5/45
Serious Adverse Events (participants affected / at risk) | 20/46 | 15/45
Other Adverse Events (participants affected / at risk) | 46/46 | 44/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niraparib + Nivolumab (Arm A) (N=46) | Niraparib + Ipilimumab (Arm B) (N=45)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (1)
Other: Acute cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Other: Passing gallbladder obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niraparib + Nivolumab (Arm A) (N=46) | Niraparib + Ipilimumab (Arm B) (N=45)
Anemia (Blood and lymphatic system disorders) | 10 (30) | 20 (41)
Palpitations (Cardiac disorders) | 0 (0) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 3 (4) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 18 (26) | 12 (15)
Constipation (Gastrointestinal disorders) | 7 (7) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 6 (9) | 12 (17)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 3 (6)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 16 (20) | 20 (25)
Vomiting (Gastrointestinal disorders) | 7 (12) | 8 (12)
Chills (General disorders) | 3 (4) | 4 (4)
Fatigue (General disorders) | 13 (18) | 26 (40)
Fever (General disorders) | 8 (10) | 10 (11)
Pain (General disorders) | 9 (13) | 4 (4)
Urinary tract infection (Infections and infestations) | 3 (4) | 1 (2)
Alanine aminotransferase increased (Investigations) | 10 (25) | 20 (30)
Alkaline phosphatase increased (Investigations) | 14 (27) | 17 (20)
Aspartate aminotransferase increased (Investigations) | 12 (33) | 22 (37)
Blood bilirubin increased (Investigations) | 7 (13) | 5 (6)
Creatinine increased (Investigations) | 5 (8) | 9 (13)
Neutrophil count decreased (Investigations) | 8 (14) | 7 (13)
Platelet count decreased (Investigations) | 18 (41) | 21 (43)
Thyroid stimulating hormone increased (Investigations) | 1 (1) | 3 (4)
Weight loss (Investigations) | 5 (5) | 6 (6)
White blood cell decreased (Investigations) | 3 (8) | 4 (11)
Anorexia (Metabolism and nutrition disorders) | 5 (6) | 6 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (6) | 5 (10)
Hypokalemia (Metabolism and nutrition disorders) | 4 (6) | 5 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 8 (8) | 11 (16)
Hyponatremia (Metabolism and nutrition disorders) | 10 (17) | 11 (17)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (5) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (11) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 8 (10)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2)
Dysgeusia (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 7 (10) | 6 (8)
Insomnia (Psychiatric disorders) | 7 (7) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 5 (7)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (8)
Other: Rash (Skin and subcutaneous tissue disorders) | 5 (7) | 5 (7)
Hot flashes (Vascular disorders) | 3 (4) | 4 (4)
Hypertension (Vascular disorders) | 6 (12) | 5 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT03404960/Prot_SAP_004.pdf
  • Informed Consent Form (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT03404960/ICF_005.pdf